CLINICAL TRIAL: NCT01642472
Title: A Phase III, Multicentre, Extension Study Investigating the Efficacy and Safety of Repeated Intermittent 3-month Courses of Open-label Administration of Ulipristal Acetate, in Subjects With Symptomatic Uterine Myomas and Heavy Uterine Bleeding
Brief Title: PGL4001 Efficacy Assessment in Reduction of Symptoms Due to Uterine Leiomyomata
Acronym: PEARLext2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PregLem SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGL11-024
Record Dates: First submitted 2012-07-10; First posted 2012-07-17 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-12

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ulipristal Acetate (PGL4001) 10mg (Experimental): Ulipristal Acetate (PGL4001)10mg daily administration
  Interventions: Drug: Ulipristal Acetate - open label

INTERVENTIONS:
Drug: Ulipristal Acetate - open label — Ulipristal Acetate (PGL4001) tablets 10mg orally daily for 3 months (84 days) for each treatment course. There are four 3-month treatment courses in this study.
  Other Names: PGL4001

SUMMARY:
This is a phase III, multicentre, long-term open-label extension of the phase III study: Pearl IIIextension (PGL09-027). During Pearl III (PGL09-026) and subsequent Pearl III extension (PGL09-027), patients have been exposed to a total of 4 cycles of daily 3month open-label treatment with ulipristal acetate 10mg before entering the proposed study Pearl extension 2 (PGL11-024).

This proposed study consists of 4 further consecutive courses of 3 months (84 days) open label ulipristal acetate 10mg once daily treatment each separated by a drug free period.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed visit F - Follow-up of Pearl III extension study (PGL09-027) - without significant deviations.
* Females of childbearing potential are advised to practice a non-hormonal method of contraception.

Exclusion Criteria:

* Subject has a history of uterus surgery (e.g. hysterectomy, myomectomy) or uterine artery embolization in Pearl III extension (PGL09-027) or afterwards that would interfere with the study assessments.
* Subject has taken or is likely to require treatment during the study with drugs that are not permitted by the study protocol.
* Subject is lactating, has a positive pregnancy test at study start or is planning a pregnancy during the course of the study.
* Subject has abnormal baseline findings, any other medical condition(s) or laboratory finding that, in the opinion of the investigator, might jeopardise the subject's safety or interfere with study evaluations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-07; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Myoma symptom control assessed with a Global Study Treatment Satisfaction Questionnaire | 9 months
  Average score of the first 3 questions.
Myoma symptom control assessed with a Global Study Treatment Satisfaction Questionnaire | 18 months
  Average score of the first 3 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Elke Bestel, Dr, Study Director — PregLem SA
Locations (16):
- Medical University Vienna, Vienna, Austria
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Gynécologie-Obstétrique,, Brussels
  - CHR de la Citadelle, Liège
  - Cliniques Universitaires UCL de Mont-Godinne, Yvoir
- Poland (8):
  - Prywatna Klinika Polozniczo-Ginekologiczna, Bialystok
  - INVICTA Sp. Z o.o., Gdansk
  - Private practice, Katowice
  - Prywatny Gabinet Lekarski Ginekologia I Poloznictwo Ultrasonografia, Lodz
  - Specjalistyczny Gabinet Ginekologiczno-Polozniczy, Lublin
  - Gabinet Lekarski Specjalistyczny "Sonus", Warsaw
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Klinika Poloznictwa, Chorob Kobiecych i Ginekologii Onkologicznej, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wrocławiu, I Katedra i Klinika Ginekologii i Położnictwa, Wroclaw
- Spain (4):
  - Hospital Universitario Vall Hebrón (Gynecology department) Edificio Maternal, Barcelona
  - Clinica Ginecologica CEOGA, Lugo
  - Private Practice, Madrid
  - HOSPITAL Universitario 12 de Octubre y Fundación de Investigación Biomédica Hospital 12 de Octubre, Madrid